CLINICAL TRIAL: NCT02577757
Title: Establishing the Language Network With Independent Component Analysis of Resting State MRI
Acronym: ICA Langage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CHU-Promoteur 2012-04
Record Dates: First submitted 2015-09-18; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Languages
Keywords: Languages network; Functional MRI
MeSH Terms: conditions — Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy volunteers (Other): achieving functional MRI
  Interventions: Device: MRI
- Eligible patients with awakened surgery (Experimental): achieving functional MRI
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI

SUMMARY:
Proceed to an analysis of sensitivity and specificity results of the fMRI language network obtained in two ways: by providing a conventional language test and independent component analysis. These two methods will be compared to the reference method what the cortical intraoperative mapping.

DETAILED DESCRIPTION:
Patients with brain tumors including malignant gliomas located in eloquent areas have long been considered inoperable because of median survival and predictable postoperative sequelae. The improved prognosis with chemoradiotherapy and surgical resection as complete as possible questioned this attitude. The goal is to operate those patients without additional disabilities. The cortical electrostimulation intraoperative mapping in awake surgery can meet the eloquent areas. Identifying with fMRI these same areas to better specify in advance the way initially and shortened the time to awake exploratory surgery which improves patient comfort. However anxiety induced by the review in a pre-operative setting, a debutante aphasia often make problematic the realization of a formal language test. The analysis in the low frequency of spontaneous oscillations of large neuronal networks can help isolate network of language at rest without particular language test at the group analysis. This methodology, however, needs to be validated at the individual level before it can be applied to pathology.

Proceed to an analysis of sensitivity and specificity results of the fMRI language network obtained in two ways: by providing a conventional language test and independent component analysis. These two methods will be compared to the reference method what the cortical intraoperative mapping.

ELIGIBILITY:
Inclusion Criteria:

* Persons major and minor.
* Having given their written consent, or whose parents have given their written consent for minors.
* Affiliated with the social security system
* All patients eligible adults in awake surgery
* Affiliated with the social security system
* patient given their written consent

Exclusion Criteria

* Contraindications to MRI
* Pregnant or breastfeeding women

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
MRI data obtained by comparing a formal language test to data obtained by a session of rest independent component analyzed in patients and volunteers | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: ARAM TER MINASSIAN, MD, Principal Investigator — UH ANGERS
Locations (1):
- CHU Angers, Angers, France